CLINICAL TRIAL: NCT05510154
Title: Impact of E-cigarette Training on Puff Patterns, Cigarette Smoking, and Health Outcomes Among Smokers With COPD
Brief Title: COPD E-cigarette Topography Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Eleanor Leavens, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147523
Record Dates: First submitted 2022-06-30; First posted 2022-08-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Tobacco Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tobacco Smoking | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: An open-label, randomized clinical trial of e-cigarette training and training dose among smokers with COPD. Smokers with COPD (n=45) stratified by e-cigarette use history (naïve vs. current use) will be randomized (1:1:1) to receive 1) brief advice to switch to e-cigarettes, 2) single session e-cigarette training, or 3) enhanced e-cigarette training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Advice (Experimental): Brief Advice involves basic e-cigarette education and advice to switch.
  Interventions: Behavioral: Brief advice
- Single Training (Experimental): Single Training is the same as Brief Advice but includes one session of real-time training on how to puff on the e-cigarette.
  Interventions: Behavioral: Single Training
- Training to Competency (Experimental): Training to Competency is the same as Single Training but includes three real-time training sessions rather than one.
  Interventions: Behavioral: Training to Competency

INTERVENTIONS:
Behavioral: Brief advice — A single, brief advice session on switching to electronic cigarettes.
  Arms: Brief Advice
Behavioral: Single Training — A single, in-depth training session on switching to electronic cigarettes.
  Arms: Single Training
Behavioral: Training to Competency — Multiple, in-depth training sessions on switching to electronic cigarettes.
  Arms: Training to Competency

SUMMARY:
This study is for people with chronic obstructive pulmonary disease (COPD) and who smoke. Investigators are trying to find out if training on e-cigarette use will help smokers switch to e-cigarettes. If training helps, how much training is needed for people to fully switch from cigarettes to e-cigarettes?

DETAILED DESCRIPTION:
Investigators are doing this study with people who smoke and have chronic obstructive pulmonary disease (COPD). Investigators are trying to find out if e-cigarettes can reduce tobacco-related harm among smokers. Investigators want to know if training on e-cigarette use will help smokers switch to e-cigarettes. If training helps, how much training is needed for people to fully switch from cigarettes to e-cigarettes? This study is an in-lab smoking study and randomized trial. The study takes place at the Main University of Kansas Medical Center (KUMC) campus in Kansas City, Kansas (KS). device. Participants will come to the lab on seven separate days. Between visits, participants will use the study e-cigarette at home. Each time participants come in, participants will fill out surveys about participants tobacco use and use the study product. Investigators will ask participants to switch to the study e-cigarette for 12 weeks during the study.

The study product is an e-cigarette device and is available for sale in the US. Participants will do a few different breathing tests where participants blow into a machine, Investigators will measure participants blood pressure and pulse, and Investigators will do a short walking test. Before three of the visits Investigators will ask participants to not smoke or use an e-cigarette for 12 hours leading up to the visit. During three of the visits, Investigators will ask participants to use the e-cigarette for 30 minutes and take two blood samples. Each visit will last about 2-4 hours. There will be a total of seven visits.

ELIGIBILITY:
Inclusion Criteria:

* Smokers:
* Diagnosed with COPD

  -≥21 years old
* Speak and understand English
* Smoke on >25 of the last 30 days for the past 3 months
* Willing to switch from cigarettes to the study e-cigarette for the duration of the study
* Have tried but failed to quit smoking in the last year
* Unwilling to make a pharmacotherapy-assisted quit attempt in the next 30 days
* Willing to complete six in-person study visits
* Willing to have blood drawn
* Have reliable transportation to attend all in-person assessments
* Have a working phone number
* Plan to remain in the Kansas City area for the full duration of the trial.

Dual users:

* Diagnosed with COPD
* ≥21 years old
* speak and understand English
* smoke on ≥15 days of the last 30 days for the past 3 months
* willing to switch from cigarettes and their own e-cigarette to the study e-cigarette for the duration of the study
* use an e-cigarette on >15 days of the last 30 days for the past 3 months
* Have tried but failed to quit smoking in the last year
* Unwilling to make a pharmacotherapy-assisted quit attempt in the next 30 days
* Willing to complete six in-person study visits
* Willing to have blood drawn
* Have reliable transportation to attend all in-person assessments
* Have a working phone number
* Plan to remain in the Kansas City area for the full duration of the trial.

Exclusion Criteria:

* Smokers:
* Use of tobacco products other than cigarettes including e-cigarettes in the past 30 days
* current use of cessation medications
* pregnant, planning to become pregnant, or breastfeeding
* recent history of cardiovascular or pulmonary events in the past 3 months
* household member current or previously enrolled in the study
* weekly use of an e-cigarette over the last 6 months
* Dual Users:
* Use of tobacco products other than cigarettes and e-cigarettes in the past 30 days
* current use of cessation medications
* pregnant, planning to become pregnant, or breastfeeding
* recent history of cardiovascular or pulmonary events in the past 3 months
* household member current or previously enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in puff duration in seconds from pre- to post-e-cigarette training | 12 weeks
  Researchers are using a puff topography device to capture real-time electronic cigarette puff and usage patterns. The electronic cigarette is attached to a device during 30-minute sessions where participants use the electronic cigarette as much or as little as they want. Researchers are measuring changes in puff duration in seconds from pre- to post-e-cigarette training/brief advice between smokers who received brief advice versus e-cigarette training (single episode and enhanced e-cigarette training arms combined). Measurements are compared from the first visit to the last visit at week 12.

SECONDARY OUTCOMES:
Complete switch to e-cigarette | 12 weeks
  Proportion of participants who completely switch e-cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Leavens, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leavens ELS, Wagener TL, Lambart L, Mayo MS, Brown L, Ellerbeck EF, Billinger SA, Comfort B, Woodward J, Sear B, Beaman S, Cox LS, Nollen NL. E-cigarette puff topography instruction to enhance switching among COPD patients who smoke. Front Public Health. 2025 Oct 2;13:1664400. doi: 10.3389/fpubh.2025.1664400. eCollection 2025. PMID 41112651

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT05510154/Prot_000.pdf
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT05510154/ICF_001.pdf